CLINICAL TRIAL: NCT06703957
Title: The Samsung Medical Center Comprehensive Cancer Center Registry from 2008 to 2023
Acronym: SCCCR08-23
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Woo Yong Lee, Chair, Samsung Medical Center
Other Study IDs: SMC cancer registry 08-23
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Neoplasm
Keywords: Cancer; Registry
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a retrospective cohort study using the Samsung Medical Center Cancer Registry, including cancer patients between 2008 and 2022.

To monitor trends in patient demographics, treatment patterns, and outcomes.

DETAILED DESCRIPTION:
All medical, administrative, and patient information is saved in an EMR system. Age at diagnosis (years), sex, body mass index, region of residence, marital status at diagnosis, employment status at diagnosis, diagnostic pathways (detected by screening, incidentally diagnosed cancer, detected by symptoms), and diagnostic method were obtained from the ERM by trained cancer registrars. Cancer types were classified based on the GLOBOCAN cancer dictionary, and the latter was the taxonomy used in "Cancer Incidence in Five Continents", and the International Association of Cancer Registries provided both of them. In this study, the cancer classification with 24 types of cancer was used for description based on the Korean National Cancer Registry annual report.

The summary staging system developed under the Surveillance, Epidemiology, and End Results (SEER) program (i.e., SEER summary staging) [12] was used to categorize the extent of tumor invasion or metastasis. Based on the 7th edition of the American Joint Committee on Cancer Staging Manual, SEER data were markedly enriched with tumor grades, invasion/metastasis status (bone, brain, lung, and liver), site-specific variables, and tumor stages.

For procedures such as genetic testing, surgery, chemotherapy and radiation therapy, clinical trial participation, and supportive care center visits, data were extracted from the DARWIN-C clinical data warehouse of Samsung Medical Center.

Trends of the hospital process included applying clinical pathways, fast track, and multi-disciplinary community were obtained from Enterprise Data Warehouse (EDW). Clinical pathways are tools used to guide evidence-based healthcare. A clinical pathway is a structured multidisciplinary care plan that details the steps in a course of treatment or care in a plan, pathway, algorithm, guideline, protocol, or other inventory of actions. The fast-track treatment system is additional tests for surgery, and decisions about surgery are all done on the first day of the visit for patients diagnosed with cancer who require surgery. Multi-disciplinary community is to bring together a group of healthcare professionals from different fields to determine patients' treatment plans. Survival status and date of death were obtained from the mortality database of the Ministry of the Interior and Safety. Overall survival (OS) was defined as the time from the date of diagnosis to death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patient who visited Samsung Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 301055 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years after cancer diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No